CLINICAL TRIAL: NCT00980980
Title: Cluster Randomized Trial of Hospitals to Assess Impact of Targeted Versus Universal
Brief Title: Cluster Randomized Trial of Hospitals to Assess Impact of Targeted Versus Universal Strategies to Reduce Methicillin-resistant Staphylococcus Aureus (MRSA) in Intensive Care Units (ICUs)
Acronym: REDUCE-MRSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); Hospital Corporation of America (Industry); University of California, Irvine (Other); Department of Population Medicine, Harvard Medical School / Harvard Pilgrim Healthcare Institute (Unknown)
Responsible Party: Principal Investigator, Richard Platt, Professor and Department Chair, Harvard Pilgrim Health Care
Allocation: Randomized | Purpose: Prevention
Other Study IDs: PH000223K; HHSA2902005003I; TO #11
Record Dates: First submitted 2009-09-19; First posted 2009-09-21 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Methicillin-resistant Staphylococcus Aureus
Keywords: MRSA infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Usual Care-Active Surveillance (No Intervention): Active Surveillance in All Adult ICUs, Contact Precautions for MRSA+
- Arm 2: Targeted Decolonization (Active Comparator): Continue Active Surveillance (AS), MRSA decolonization based on AS, Continue Contact Precautions for MRSA+
  Interventions: Drug: Chlorhexidine bath and nasal mupirocin
- Arm 3: Universal Decolonization (Active Comparator): Chlorhexidine bath and nasal mupirocin for all, Discontinuation of Active Surveillance, Continuation of Contact Precautions for MRSA+
  Interventions: Drug: Chlorhexidine bath and nasal mupirocin

INTERVENTIONS:
Drug: Chlorhexidine bath and nasal mupirocin — The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths , plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
  Arms: Arm 2: Targeted Decolonization; Arm 3: Universal Decolonization

SUMMARY:
The Randomized Evaluation of Decolonization versus Universal Clearance to Eliminate MRSA (REDUCE MRSA) Trial is a cluster randomized trial of the comparative effectiveness of three strategies to prevent methicillin-resistant Staphylococcus aureus (MRSA) in intensive care units. The three strategies to be evaluated are:

* screening on admission followed by isolation of MRSA+ patients
* screening on admission followed by isolation and decolonization of MRSA+ patients
* universal decolonization on admission with no screening. The decolonization regimen involves bathing with chlorhexidine plus intra-nasal application of mupirocin. The main outcome will be MRSA+ clinical cultures.

The study is a partnership between the CDC, the CDC Prevention Epicenters, and the Hospital Corporation of America.

DETAILED DESCRIPTION:
Baseline data involving 12 months of data for participating hospitals (July 2008 - June 2009) was collected prior to randomization to account for size and ICU baseline prevalence of MRSA in randomization scheme. Randomization occurred at the hospital level.

Eligibility survey was conducted to determine exclusion criteria.

As of May 2010, enrollment has been closed. 45 hospitals were randomized, but two were found to meet exclusion criteria and were excluded. As-randomized (or as-assigned) analysis included 43 hospitals, representing 74 ICUs. Individual (patient-level) subject enrollment during intervention is 74,256.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include all HCA hospitals that reside in US states where physicians do NOT routinely prescribe decolonization for MRSA + ICU patients.

Exclusion Criteria:

* Exclusion criteria will include hospitals where ICU physicians often prescribe decolonization for MRSA+ ICU patients.
* Dedicated burn ICUs will also be excluded due to the inability to perform routine bathing.
* Finally, since the intent is to assess the intervention in adult ICUs, pediatric hospitals will be excluded although patients <13 years old that are admitted to participating adult ICUs will be included in the unit-based intervention.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74256 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Platt, MD, MS, Principal Investigator — Department of Population Medicine, Harvard Medical School / Harvard Pilgrim Healthcare Institute; Edward Septimus, MD, Principal Investigator — Hospital Corporation of America; Susan Huang, MD MPH, Principal Investigator — University of California, Irvine
Locations (42):
- United States (42):
  - Alaska Regional, Anchorage, Alaska
  - Los Robles Hosp & Med Ctr, Thousand Oaks, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Blake Medical Center, Brandenton, Florida
  - Brandon Hospital, Brandon, Florida
  - Columbia Hosp Corp S Broward (Westside), Fort Lauderdale, Florida
  - Palms West Hospital, Fort Lauderdale, Florida
  - Plantation General, Fort Lauderdale, Florida
  - Regional Med Cr Bayonet Point, Hudson, Florida
  - Largo Medical Center, Largo, Florida
  - Community Hospital, New Port Richey, Florida
  - Orange Park Med Ctr, Orange Park, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Doctors Hospital of Sarasota, Sarasota, Florida
  - South Bay Hospital, Sun City Center, Florida
  - Capital Regional Med Ctr, Tallahassee, Florida
  - Coliseum (Macon) Northside, Macon, Georgia
  - Coliseum Medical Center, Macon, Georgia
  - Cartersville Medical Center, Tucker, Georgia
  - Eastern Idaho Reg Med Ctr, Idaho Falls, Idaho
  - Garden Park Medical Center, Gulfport, Mississippi
  - Lee's Summit Medical Center, Kansas City, Missouri
  - Menorah Medical Center, Kansas City, Missouri
  - Overland Park Regional Hospital, Kansas City, Missouri
  - Research Belton Hospital, Kansas City, Missouri
  - Moutainview Medical Center, Las Vegas, Nevada
  - Parkland Medical Center, Derry, New Hampshire
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Parkridge Medical Center, Chattanooga, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Stonecrest, Smyrna, Tennessee
  - St. David's Medical Center, Austin, Texas
  - Del Sol Medical Center, El Paso, Texas
  - Las Palmas Medical Center, El Paso, Texas
  - Medical Center of Plano, Plano, Texas
  - Methodist Hospital, San Antonio, Texas
  - Clear Lake Regional, Webster, Texas
  - Montgomery Regional Hospital, Blacksburg, Virginia
  - Columbia Alleghany Regional Hospital, Low Moor, Virginia
  - Pulaski Community Hospital, Pulaski, Virginia
  - Chippenham Johnston Willis, Richmond, Virginia

REFERENCES:
- [Background] Platt R, Takvorian SU, Septimus E, Hickok J, Moody J, Perlin J, Jernigan JA, Kleinman K, Huang SS. Cluster randomized trials in comparative effectiveness research: randomizing hospitals to test methods for prevention of healthcare-associated infections. Med Care. 2010 Jun;48(6 Suppl):S52-7. doi: 10.1097/MLR.0b013e3181dbebcf. PMID 20473200
- [Background] Huang SS, Septimus E, Platt R. Targeted decolonization to prevent ICU infections. N Engl J Med. 2013 Oct 10;369(15):1470-1. doi: 10.1056/NEJMc1309704. No abstract available. PMID 24106942
- [Result] Huang SS, Septimus E, Kleinman K, Moody J, Hickok J, Avery TR, Lankiewicz J, Gombosev A, Terpstra L, Hartford F, Hayden MK, Jernigan JA, Weinstein RA, Fraser VJ, Haffenreffer K, Cui E, Kaganov RE, Lolans K, Perlin JB, Platt R; CDC Prevention Epicenters Program; AHRQ DECIDE Network and Healthcare-Associated Infections Program. Targeted versus universal decolonization to prevent ICU infection. N Engl J Med. 2013 Jun 13;368(24):2255-65. doi: 10.1056/NEJMoa1207290. Epub 2013 May 29. PMID 23718152
- See also: NEJM Study Results Publication — http://www.nejm.org/doi/full/10.1056/NEJMoa1207290
- See also: AHRQ Toolkit: Universal ICU Decolonization: An Enhanced Protocol — http://www.ahrq.gov/professionals/systems/hospital/universal_icu_decolonization/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 out of 165 Hospital Corporation of America (HCA) hospitals were recruited for this trial of adult ICUs. There was a 12-month baseline period from January 1 through December 31, 2009; a phase-in period from January 1 through April 7, 2010; and an 18-month intervention period from April 8, 2010 through September 30, 2011.
Pre-assignment Details: 74,256 patients were involved in the intervention period among adult ICUs from the 43 participating hospitals. Routinely collected information for about 48,390 individuals cared for during the baseline period was used for comparison to the experience of the patients in all three arms of the Intervention period.
Groups:
- Arm 2: Targeted Decolonization: Continue Active Surveillance (AS), MRSA decolonization based on AS, Continue Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of baths with 2% chlorhexidine cloths plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
- Arm 3: Universal Decolonization: Chlorhexidine bath and nasal mupirocin for all, Discontinuation of Active Surveillance , Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
Period: Overall Study
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Started | 16 | 14 | 13
Completed | 16 | 13 | 13
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Hospital | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 'Number of Participant' totals reflect total Baseline and Intervention participants combined. 45 hospitals were randomized to a study group, 2 dropped due to exclusion criteria, 43 began the assigned intervention. 1 hospital withdrew during the intervention and was included in as-assigned analyses.
Groups:
- Arm 2: Targeted Decolonization: Continue Active Surveillance (AS), MRSA decolonization based on AS, Continue Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
- Arm 3: Universal Decolonization: Chlorhexidine bath and nasal mupirocin for all, Discontinuation of Active Surveillance, Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
- Total: Total of all reporting groups
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization | Total
Number analyzed (Participants) | 39296 | 39970 | 43380 | 122646
Age, Continuous [Median (Inter-Quartile Range); unit: Years]
  Baseline Age | 65 [52 to 77] | 66 [53 to 77] | 65 [51 to 77] | 65 [52 to 77]
  Intervention Age | 65 [52 to 77] | 66 [53 to 77] | 65 [52 to 77] | 65 [52 to 77]
Sex/Gender, Customized [Number; unit: participants] — Proportion of female study participants, during baseline and intervention study phases.
  participants
    Females - Baseline | 7465 | 7183 | 8314 | 22962
    Males - Baseline | 8351 | 8035 | 9042 | 25428
    Females - Intervention | 11176 | 11683 | 12361 | 35220
    Males - Intervention | 12304 | 13069 | 13663 | 39036
Overall Number of Participants, by Phase [Number; unit: Admissions] — This table reflects number of admissions with an ICU stay during the Baseline and Intervention periods, separately. Please note that the table above, "Overall Number of Baseline Participants" reflects the total number of participants for which baseline characteristics were measured, across Baseline and Intervention phases combined.
  Admissions
    Baseline Participants | 15816 | 15218 | 17356 | 48390
    Intervention Participants | 23480 | 24752 | 26024 | 74256

OUTCOME MEASURES:

1. Primary Outcome: Main Outcome: Patients With Nosocomial MRSA Clinical Cultures
Description: Hazard ratio for ICU-attributable MRSA+ clinical cultures comparing Baseline to Intervention period, by Arm, accounting for clustering by hospital.
Time Frame: The 30-month time frame represents 12-month baseline and 18-month intervention periods. During these time periods, outcomes are defined as events occurring during attributed ICU time: from day 3 of the ICU stay until 2 days after ICU discharge.
Population: The total number of participants analyzed included the table reflects the combined total of baseline and intervention participants, for each arm.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Arm 2: Targeted Decolonization: Continue Active Surveillance (AS), MRSA decolonization based on AS, Continue Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths, plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
- Arm 3: Universal Decolonization: Chlorhexidine bath and nasal mupirocin for all, Discontinuation of Active Surveillance , Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths, plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 39296 | 39970 | 43380
hazard ratio | 0.92 [0.77 to 1.10] | 0.75 [0.63 to 0.89] | 0.63 [0.52 to 0.75]
Statistical Analysis 1: Comparison: Arm 1: Usual Care-Active Surveillance vs Arm 2: Targeted Decolonization vs Arm 3: Universal Decolonization; Test type: Superiority or Other; p = 0.01, Proportional-hazards models; Proportional-hazards models with shared frailties accounted for clustering within hospitals

2. Secondary Outcome: MRSA Bloodstream Infection
Description: Hazard ratio for ICU-attributable MRSA+ blood cultures comparing Baseline to Intervention period, by Arm, accounting for clustering by hospital.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Arm 3: Universal Decolonization: Chlorhexidine bath and nasal mupirocin for all, Discontinuation of Active Surveillance, Contact Precautions for MRSA+
  Chlorhexidine bath and nasal mupirocin: The intervention / decolonization regimen will consist of the most commonly used topical regimen in the US - a combination of daily baths with 2% chlorhexidine cloths, plus 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily)
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 39296 | 39970 | 43380
hazard ratio | 1.23 [0.82 to 1.85] | 1.23 [0.80 to 1.90] | 0.72 [0.48 to 1.08]

3. Secondary Outcome: ICU-attributable All-pathogen Bloodstream Infection
Description: Hazard ratio for ICU-attributable positive blood culture from any pathogen, comparing Baseline to Intervention period, by Arm, accounting for clustering by hospital.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 39296 | 39970 | 43380
Hazard ratio | 0.99 [0.84 to 1.16] | 0.78 [0.66 to 0.91] | 0.56 [0.49 to 0.65]

4. Secondary Outcome: Intervention Impact on Healthcare Costs
Description: Costs (in dollars) per 1000 ICU-admissions associated with 3 ICU strategies to reduce ICU Bloodstream infection (BSI), (Arms 1-3).
Time Frame: 12-month period
Population: Annual adult ICU admissions per hospital, over the course of 1 year.
Measure: Number; unit: Dollars per 1000 ICU-admissions
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 1000 | 1000 | 1000
Dollars per 1000 ICU-admissions
  Cost of MRSA screening tests | 9,120 | 9,120 | 0
  Cost of contact precautions | 69,010 | 68,830 | 24,890
  Cost of decolonization | 0 | 4,679 | 36,500
  ICU costs (not including intervention costs) | 19,320,000 | 19,250,000 | 19,170,000

5. Secondary Outcome: Blood Culture Contamination Rates
Description: Odds ratio for ICU-attributable blood culture contamination rates, comparing Baseline to Intervention period across Arms, accounting for clustering by hospital.
Time Frame: 24-month time frame for this analysis represents a 6-month baseline and 18-month intervention period.
Population: The number of participants analyzed reflects the combined total of baseline and intervention admissions, with an ICU stay and a blood draw set, for each arm.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 4154 | 4141 | 4982
Odds Ratio
  As randomized, unadjusted | 0.74 [0.58 to 0.94] | 0.94 [0.72 to 1.23] | 0.56 [0.44 to 0.71]
  As randomized, adjusted | 0.73 [0.57 to 0.94] | 0.93 [0.7 to 1.22] | 0.55 [0.43 to 0.71]

6. Secondary Outcome: Intervention Impact on Bacteriuria and Candiduria
Description: Proportional hazard ratio for as-randomized, unadjusted, ICU-attributable bacteriuria, comparing Baseline to Intervention period across Arms, accounting for clustering by hospital. High-level bacteriuria is defined as ≥50,000 CFU/mL, high-level candiduria is defined as ≥50,000 CFU/mL.
Time Frame: 30-month time frame represents 12-month baseline and 18-month intervention periods.
Population: The number of participants analyzed reflects the combined total of baseline and intervention admissions with an ICU stay, for each arm.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 39296 | 39970 | 43380
Hazard Ratio
  High-level bacteriuria (all patients) | 1.02 [0.88 to 1.18] | 0.88 [0.76 to 1.02] | 0.87 [0.77 to 1.00]
  High-level bacteriuria (women) | 0.97 [0.80 to 1.17] | 0.83 [0.70 to 1.00] | 0.93 [0.79 to 1.09]
  High-level bacteriuria (men) | 1.09 [0.85 to 1.40] | 1.01 [0.79 to 1.29] | .78 [.63 to .98]
  High-level candiduria (all patients) | 1.14 [.95 to 1.37] | .99 [.83 to 1.18] | .83 [.70 to .99]
  High-level candiduria (women) | 1.09 [.88 to 1.36] | 1.00 [.81 to 1.24] | .94 [.76 to 1.16]
  High-level candiduria (men) | 1.21 [.88 to 1.68] | 1.01 [.73 to 1.39] | .63 [.45 to .89]
  Any bacteriuria (all patients) | .95 [.84 to 1.09] | .92 [.8 to 1.04] | .86 [.77 to .97]
  Any bacteriuria (women) | .91 [.77 to 1.08] | .86 [.73 to 1.01] | .95 [.82 to 1.10]
  Any bacteriuria (men) | 1.01 [.81 to 1.25] | 1.04 [.83 to 1.3] | .74 [0.61 to .9]

7. Secondary Outcome: Intervention Impact on Mupirocin Susceptibility of MRSA Isolates
Description: Odds ratio for MRSA+ isolates from ICU patients expressing low-level mupirocin resistance (LLMR) and high-level mupirocin resistance (HLMR), comparing baseline to intervention period across arms, accounting for clustering by hospital.
Time Frame: 25-month time frame represents 7-month baseline and 18-month intervention periods
Population: The total number of participants analyzed reflects the combined total of baseline and intervention participants during the outcome time frame, for each arm. The total number of units analyzed reflects the combined total of MRSA+ isolates collected from ICU patients during baseline and intervention phase, for each arm.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Units Other Than Participants: MRSA+ isolates
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 29643 | 28297 | 32601
Number analyzed (MRSA+ isolates) | 1303 | 1460 | 410
Odds Ratio
  Clinical MRSA: LLMR | 1.0 [0.22 to 4.85] | 1.4 [0.34 to 6.14] | 0.5 [0.1 to 2.14]
  Clinical MRSA: HLMR | 0.8 [0.11 to 5.68] | 0.9 [0.15 to 5.44] | 0.7 [0.16 to 3.01]
  ICU-attributable MRSA: LLMR | 1.7 [0.37 to 7.55] | 0.4 [0.01 to 99] | 0.7 [0.10 to 4.64]
  ICU-attributable MRSA: HLMR | 1.5 [0.25 to 9.02] | 0.7 [0.09 to 5.06] | 1.4 [0.134 to 15.63]

8. Secondary Outcome: Intervention Impact on Chlorhexidine Susceptibility of MRSA Isolates
Description: Frequency of MRSA+ isolates from ICU patients with reduced susceptibility to chlorhexidine (CHG) (MIC >4 μg/ml), comparing baseline to intervention period across arms, accounting for clustering by hospital.
Time Frame: 25-month time frame represents 7-month baseline and 18-month intervention periods
Population: as for outcome 7
Measure: Number; unit: MRSA isolates non-susceptible to CHG
Units Other Than Participants: MRSA+ isolates
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Number analyzed (Participants) | 29643 | 28297 | 32601
Number analyzed (MRSA+ isolates) | 1303 | 1460 | 410
MRSA isolates non-susceptible to CHG | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse event monitoring and reporting occurred during intervention only, as decolonizing agents were not used during the baseline period.
Groups:
- Arm 1: Usual Care-Active Surveillance: Active Surveillance in All Adult ICUs Contact Precautions for MRSA+
Arm/Group | Arm 1: Usual Care-Active Surveillance | Arm 2: Targeted Decolonization | Arm 3: Universal Decolonization
Serious Adverse Events (participants affected / at risk) | 0/23480 | 0/24752 | 0/26024
Other Adverse Events (participants affected / at risk) | 0/23480 | 2/24752 | 5/26024
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Usual Care-Active Surveillance (N=23480) | Arm 2: Targeted Decolonization (N=24752) | Arm 3: Universal Decolonization (N=26024)
Mild (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (5) — A mild adverse event included any criteria less than moderate
Moderate (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) — A moderate adverse event included any moderate erythema, scaling or blistering that involves >30% body surface area
Severe (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) — A severe adverse event included any severe erythema, scaling or blistering that involves >30% body surface area

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No